CLINICAL TRIAL: NCT06120257
Title: Flexible Ureteroscopy , Extracorporeal Shock Wave Lithotripsy and Mini Percutaneous Nephrolithotomy for Management of Lower Pole Renal Hard Stones ≤2 cm: Prospective Comparative Study
Brief Title: Management of Lower Pole Renal Hard Stones ≤2 cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsayed Abdelhalim Elsayed (Other)
Responsible Party: Sponsor-Investigator, Elsayed Abdelhalim Elsayed, Principal Investigator, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-69
Record Dates: First submitted 2023-10-22; First posted 2023-11-07 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Renal Stones
Keywords: Hard stones
MeSH Terms: conditions — Nephrolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A :Flexible ureteroscope group (Active Comparator): Flexible ureteroscope (F-URS) group underwent holmium laser lithotripsy using flexible ureteroscopy (Boston® scientific (lithovue)
  Interventions: Procedure: lithotripsy using Flexible ureteroscope
- Group B : extracorporeal shock wave lithotripsy (ESWL) group (Active Comparator): extracorporeal shock wave lithotripsy (ESWL) group underwent electromagnetic extracorporeal shock wave lithotripsy (STORZ® MEDICAL Modulith SLX-F2 FD21, Germany)
  Interventions: Procedure: extracorporeal shock wave lithotripsy (ESWL)
- Group C : Mini perc group (Active Comparator): Mini perc group underwent holmium laser lithotripsy using Karl® Storz MIP set.
  Interventions: Procedure: holmium laser lithotripsy using Karl® Storz MIP set

INTERVENTIONS:
Procedure: lithotripsy using Flexible ureteroscope — using Flexible ureteroscope and holmium laser lithotripsy to get high stone clearance rate
  Arms: Group A :Flexible ureteroscope group
Procedure: extracorporeal shock wave lithotripsy (ESWL) — using extracorporeal shock wave lithotripsy (ESWL) to get high stone clearance rate
  Arms: Group B : extracorporeal shock wave lithotripsy (ESWL) group
Procedure: holmium laser lithotripsy using Karl® Storz MIP set — using holmium laser lithotripsy using Karl® Storz MIP set to get high stone clearance rate
  Arms: Group C : Mini perc group

SUMMARY:
The study has been conducted in Urology department at Kafrelsheikh University Hospital between March 2022 to March 2023. informed consent was taken from eligible patients and were randomized into three groups, Group A :Flexible ureteroscope (F-URS) group underwent holmium laser lithotripsy using flexible ureteroscopy (Boston® scientific (lithovue) while, Group B : extracorporeal shock wave lithotripsy (ESWL) group underwent electromagnetic extracorporeal shock wave lithotripsy (STORZ® MEDICAL Modulith SLX-F2 FD21, Germany) .Group C : Mini perc group underwent holmium laser lithotripsy using Karl® Storz MIP set.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient older than 18 years.
* single renal stone.
* medium sized Stone up to 2.0 cm .
* Do novo
* Stone in lower calyceal stone
* Hard stone

Exclusion Criteria:

* • multiple renal stones

  * stone size > 2 cm
  * age group < 18
  * solitary kidney
  * Patients with BMI > 40 kg/m2
  * bleeding disorders
  * anatomical renal abnormalities
  * Obstruction distal to the stone.
  * Musculoskeletal deformities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
stone free rate | after two weeks from primary procedure
  no stone residual fragments or asymptomatic insignificant residual fragments less than or equal to 4 mm during patients follow up two weeks.

SECONDARY OUTCOMES:
assess operative time. | during the procedure
  assess operative time.in minutes
visual analog scale | immediately after the surgery
  Patient self dependent to assess degree of own pain, consists of a 10cm line, with two end points representing 0 minimum score('no pain') and 10 maximum score('pain as bad as it could possibly be').higher scores mean a worse outcome.
Radiation time | during the procedure
  Time of patient exposure for radiation in minutes
Post operative complication | Up to 48 hours
  Complication may occur post operative complication like fever, sever pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zeinelabden KM, Abdelhalim E, Galal M, Abdelbaky T, Nabeeh H. Flexible ureteroscopy, extracorporeal shock wave lithotripsy and mini percutaneous nephrolithotomy for management of lower pole renal hard stones </= 2 cm: a prospective randomized study. BMC Urol. 2024 Dec 30;24(1):288. doi: 10.1186/s12894-024-01644-z. PMID 39736616